CLINICAL TRIAL: NCT00180024
Title: Characterization of Vascular Effects of Angiotensin II in Dorsal Human Hand Veins.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: IKPD 01-02
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Healthy Subjects
Keywords: AT1-receptor; AT2-receptor; human pharmacology
MeSH Terms: interventions — Irbesartan; Pharmaceutical Preparations

INTERVENTIONS:
Drug: irbesartan (drug)

SUMMARY:
The hypothesis is tested that stimulation with angiotensin II after blockade of the AT1-receptor results in venodilation in human healthy subjects in vivo.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* any relevant disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2002-01; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, Study Chair — Institute of Clinical Pharmacology
Locations (1):
- Institute of Clinical Pharmacology, Medical Faculty, University of Technology, Dresden, Germany